CLINICAL TRIAL: NCT03071263
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group Study of Patiromer for the Enablement of Spironolactone Use for Blood Pressure Control in Patients With Resistant Hypertension and Chronic Kidney Disease
Brief Title: Spironolactone With Patiromer in the Treatment of Resistant Hypertension in Chronic Kidney Disease
Acronym: AMBER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Relypsa, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLY5016-207; 2016-002657-38 (EudraCT Number)
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Hyperkalemia; Resistant Hypertension
Keywords: Treatment of Hyperkalemia; Hyperkalemia; Potassium; Chronic Kidney Disease; Hypertension; Resistant Hypertension; Spironolactone
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic; Hypertension | interventions — patiromer; Suspensions; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - Patiromer (Experimental): spironolactone + blinded patiromer
  Interventions: Drug: Patiromer; Drug: Spironolactone
- Group 2 - Placebo (Experimental): spironolactone + blinded placebo
  Interventions: Drug: Placebo; Drug: Spironolactone

INTERVENTIONS:
Drug: Patiromer — 2 packets/day starting dose, administered orally
  Other Names: Veltassa; RLY5016 for Oral Suspension; Patiromer for Oral Suspension
  Arms: Group 1 - Patiromer
Drug: Placebo — 2 packets/day starting dose, administered orally
  Arms: Group 2 - Placebo
Drug: Spironolactone — 25 mg tablet/day starting dose, administered orally

SUMMARY:
The purpose of this study is to determine if patiromer treatment in chronic kidney disease (CKD) subjects receiving spironolactone for the treatment of resistant hypertension will result in more persistent use of spironolactone through prevention of hyperkalemia and lead to improved blood pressure control compared with treatment with spironolactone alone (placebo).

DETAILED DESCRIPTION:
Approximately 290 eligible participants with [chronic kidney disease (CKD) on stable doses of medication] will be randomly assigned to receive a patiromer or placebo starting dose of two packets a day, once a day.

All eligible participants will undergo a screening/run-in period (up to 4 weeks) to determine eligibility for study entry. Eligible participants will be randomized and treated for 12 weeks (Treatment Period) and followed for 2 weeks after completing the patiromer or placebo treatment. There are 8 planned clinic visits during the Treatment Period and one planned visit two weeks after the last dose of patiromer or placebo (Follow-up Period).

The dose of patiromer or placebo may be increased or decreased (titrated) based on participants' individual potassium response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Taking at least three medications for blood pressure (one a diuretic)
* Uncontrolled high blood pressure
* Abnormal kidney function (with-eGFR, a measure of kidney function, of 25 - ≤ 45 mL/min/1.73m2
* Normal Blood serum Potassium in a specific range (4.3 - 5.1 mEq/L)

Exclusion Criteria:

* History of untreated known causes of high blood pressure, excluding kidney disease (not CKD)
* Inability to measure BP
* Not taking high blood pressure medications as prescribed medications
* Recent change in renal function (in the past 3 months) which has required hospitalization or dialysis
* Renal transplant
* History of cancer within past 12 months
* Recent cardiovascular event with last 3 months
* Clinically significant abnormalities of heart rhythm (ventricular arrhythmia or atrial fibrillation with uncontrolled heart rate)
* Inability to take study medication
* Alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director or VP Clinical Development, Study Director — Relypsa, Inc.
Locations (40):
- United States (3):
  - Investigator Site 1012, Hollywood, Florida
  - Investigator Site 1023, Miami Lakes, Florida
  - Investigator Site 1022, Chicago, Illinois
- Investigator Site 1402, Sofia, Bulgaria
- Croatia (4):
  - Investiagor Site 2205, Zagreb
  - Investigator Site 2201, Zagreb
  - Investigator Site 2202, Zagreb
  - Investigator Site 2203, Zagreb
- Georgia (12):
  - Investigator Site 3806, Tbilisi
  - Investigator Site 3811, Tbilisi
  - Investigator Site 3802, Tbilisi
  - Investigator Site 3801, Tbilisi
  - Investigator Site 3804, Tbilisi
  - Investigator Site 3805, Tbilisi
  - Investigator Site 3807, Tbilisi
  - Investigator Site 3808, Tbilisi
  - Investigator Site 3810, Tbilisi
  - Investigator Site 3812, Tbilisi
  - Investigator Site 3813, Tbilisi
  - Investigator Site 3809, Tbilisi
- Investigator Site 4202, Göttingen, Germany
- Hungary (8):
  - Investigator Site 4607, Balatonfüred
  - Investigator Site 4606, Budapest
  - Investigator Site 4611, Debrecen
  - Investigator Site 4601, Hatvan
  - Investigator Site 4605, Kistarcsa
  - Investigator Site 4602, Miskolc
  - Investigator Site 4610, Miskolc
  - Investigator Site 4608, Mosonmagyaróvár
- Investigator Site 7403, Johannesburg, South Africa
- Ukraine (8):
  - Investiagor Site 7809, Kharkiv
  - Investigator Site 7803, Kharkiv
  - Investigator Site 7808, Kharkiv
  - Investigator Site 7802, Kharkiv
  - Investigator Site 7805, Kiev
  - Investigator Site 7801, Kiev
  - Investigator Site 7804, Zaporizhzhia
  - Investigator Site 7807, Zaporizhzhia
- United Kingdom (2):
  - Investigator Site 8202, Leicester
  - Investigator Site 8205, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal R, Rossignol P, Budden J, Mayo MR, Arthur S, Williams B, White WB. Patiromer and Spironolactone in Resistant Hypertension and Advanced CKD: Analysis of the Randomized AMBER Trial. Kidney360. 2021 Jan 15;2(3):425-434. doi: 10.34067/KID.0006782020. eCollection 2021 Mar 25. PMID 35369022
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430
- [Derived] Agarwal R, Rossignol P, Romero A, Garza D, Mayo MR, Warren S, Ma J, White WB, Williams B. Patiromer versus placebo to enable spironolactone use in patients with resistant hypertension and chronic kidney disease (AMBER): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet. 2019 Oct 26;394(10208):1540-1550. doi: 10.1016/S0140-6736(19)32135-X. Epub 2019 Sep 15. PMID 31533906
- [Derived] Agarwal R, Rossignol P, Garza D, Mayo MR, Warren S, Arthur S, Romero A, White WB, Williams B. Patiromer to Enable Spironolactone Use in the Treatment of Patients with Resistant Hypertension and Chronic Kidney Disease: Rationale and Design of the AMBER Study. Am J Nephrol. 2018;48(3):172-180. doi: 10.1159/000492622. Epub 2018 Sep 3. PMID 30176673

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Started | 147 | 148
Completed | 144 | 141
Not Completed | 3 | 7
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Participant moved to another city | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo | Total
Number analyzed (Participants) | 147 | 148 | 295
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 44 | 93
  >=65 years | 98 | 104 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (12.24) | 68.5 (11.13) | 68.1 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 71 | 142
  Male | 76 | 77 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 16 | 23
  Not Hispanic or Latino | 140 | 131 | 271
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 145 | 145 | 290
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Baseline central laboratory serum potassium [Count of Participants; unit: Participants]
  Baseline serum potassium <4.3 mEq/L | 7 | 17 | 24
  Baseline serum potassium 4.3-<4.7 mEq/L | 55 | 52 | 107
  Baseline serum potassium 4.7-5.1 mEq/L | 65 | 65 | 130
  Baseline serum potassium >5.1 mEq/L | 20 | 14 | 34
Baseline eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] — eGFR = Estimated glomerular filtration range
  mL/min/1.73m^2 | 35.37 (7.274) | 36.08 (7.597) | 35.73 (7.434)
Systolic blood pressure as measured using automated office blood pressure device (AOBP SBP) [Mean (Standard Deviation); unit: mmHg] | 143.3 (6.48) | 144.9 (7.01) | 144.1 (6.79)
Antihypertensive Medications at Baseline [Count of Participants; unit: Participants] — Antihypertensive Medications at Baseline by Preferred Drug Name for ≥10% of the total participants.
  Therapeutic Subgroup:
  * Agents Acting on the Renin-Angiotensin System (Perindopril, Valsartan, Losartan).
  * Diuretics (Indapamide, Hydrochlorothiazide, Furosemide, Torasemide)
  * Calcium Channel Blockers (Amlodipine, Lercanidipine)
  * Beta Blocking Agents (Bisoprolol, Nebivolol)
  * Other antihypertensives (Moxonidine, Rilmenidine, Doxazosin, Clonidine, Prazosin, Urapidil, Dihydralazine, Hydralazine, Reserpine, Terazosin)
  Participants
    Perindopril | 54 | 51 | 105
    Valsartan | 38 | 27 | 65
    Losartan | 20 | 26 | 46
    Indapamide | 62 | 58 | 120
    Hydrochlorothiazide | 52 | 60 | 112
    Furosemide | 26 | 17 | 43
    Torasemide | 15 | 17 | 32
    Amlodipine | 74 | 86 | 160
    Lercanidipine | 18 | 15 | 33
    Bisoprolol | 34 | 43 | 77
    Nebivolol | 26 | 19 | 45
    Other antihypertensives | 40 | 31 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Remaining on Spironolactone at Week 12
Description: The proportion of subjects remaining on spironolactone at Week 12 will be compared between treatment groups (spironolactone/patiromer versus spironolactone/placebo). Subjects who discontinued from the study early or discontinued study spironolactone prior to Week 12, for any reason, were considered as not having remained on spironolactone until Week 12.
Time Frame: At week 12
Population: Intent-to-Treat population (ITT): The ITT population included all participants who were randomized and who took at least 1 dose of spironolactone and at least 1 dose of patiromer/placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 147 | 148
Participants | 126 | 98
Statistical Analysis 1: Comparison: Group 1 - Patiromer vs Group 2 - Placebo; A sample size of 280 subjects has 90% power to detect a difference between treatment groups of 20% or more in the proportion of subjects remaining on spironolactone at Week 12, at α = 0.05; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — α-level 0.05. Stratified by baseline potassium category (4.3-<4.7 mEq/L or 4.7-5.1 mEq/L) and history of Type 1 or Type 2 diabetes mellitus (Yes or No) as randomized

2. Secondary Outcome: Change in AOBP SBP From Baseline to Week 12 or Last Available AOBP SBP Prior to Addition of Any New BP Medications or Increase From Any Baseline BP Medications
Description: AOBP: Automated Office Blood Pressure SBP: Systolic Blood Pressure BP: Blood Pressure
Time Frame: From baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 144 | 141
mmHg | -11.3 (14.11) | -11.0 (15.34)
Statistical Analysis 1: Comparison: Group 1 - Patiromer vs Group 2 - Placebo; Test type: Superiority; p = 0.5757, ANCOVA — Baseline AOBP SBP as a covariate and treatment group, baseline serum potassium (K+ 4.3-<4.7 or 4.7-5.1 mEq/L), and history of Type 1 or Type 2 diabetes mellitus (Yes or No) as factors in the model

3. Other Pre Specified Outcome: Change in AOBP SBP From Baseline to Week 12 Regardless of Increase in Antihypertensives
Description: AOBP SBP: Automated Office Systolic Blood Pressure
Time Frame: From baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 144 | 141
mmHg | -11.3 (14.11) | -11.2 (15.04)
Statistical Analysis 1: Comparison: Group 1 - Patiromer vs Group 2 - Placebo; The p-value is from a test comparing the difference between two groups in the mean change in AOBP SBP from baseline; Test type: Superiority; p = 0.6367, ANCOVA — Baseline AOBP SBP as a covariate and treatment group, baseline serum potassium (K+ 4.3-<4.7 or 4.7-5.1 mEq/L), and history of Type 1 or Type 2 diabetes mellitus as factors in the model

4. Other Pre Specified Outcome: Central Serum Potassium Change From Baseline to Week 12 by Baseline Serum Potassium Category
Description: The two baseline potassium subgroups, 4.3-<4.7 mEq/L versus 4.7-5.1 mEq/L, are based on central laboratory data.
  If a participant's serum potassium result at baseline was not in one of the two subgroups reported below, the participant's potassium stratum at randomization was used. Therefore, participants with BCSP <4.3 mEq/L or >5.1 mEq/L at baseline (Day 0) have been classified according to their serum potassium values at the Screening period.
Time Frame: From baseline to Week 12
Population: Intent-to-Treat population (ITT): The ITT population included all participants who were randomized and who took at least 1 dose of spironolactone and at least 1 dose of patiromer/placebo.
  Table depicts those participants with values at Baseline and Week 12. Those participants with no available results at W12 were not included in the table below.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 144 | 140
mEq/L
  Baseline Central Serum Potassium 4.3-<4.7 mEq/L: number analyzed (Participants) | 62 | 64
  Baseline Central Serum Potassium 4.3-<4.7 mEq/L | 0.16 (0.468) | 0.40 (0.494)
  Baseline Central Serum Potassium 4.7-<5.1 mEq/L: number analyzed (Participants) | 82 | 76
  Baseline Central Serum Potassium 4.7-<5.1 mEq/L | -0.09 (0.442) | 0.03 (0.468)
  Overall | 0.02 (0.469) | 0.20 (0.514)

5. Other Pre Specified Outcome: Participants With Central Serum Potassium <5.5 mEq/L Over Time
Description: Baseline Central Serum Potassium: BCSP.
  The symbols > and ≤ included in the row titles are used to indicate the time interval [">Week1 and ≤Week2" meaning from day 8 until day 14 (included)].
  If a participant's serum potassium result at baseline was not in one of the two subgroups reported below, the participant's potassium stratum at randomization was used. Therefore, participants with BCSP <4.3 mEq/L or >5.1 mEq/L at baseline (Day 0) have been classified according to their serum potassium values at the Screening period.
Time Frame: From baseline to Week 12
Population: Intent-to-Treat population (ITT): The ITT population included all participants who were randomized and who took at least 1 dose of spironolactone and at least 1 dose of patiromer/placebo.
  Table depicts those participants with values at mentioned time frame. Those participants with no available results were not included in the table below.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 147 | 148
Participants
  BCSP 4.3-<4.7mEq/L: ≤Week1: number analyzed (Participants) | 63 | 66
  BCSP 4.3-<4.7mEq/L: ≤Week1 | 60 | 62
  BCSP 4.3-<4.7mEq/L: >Week1 and ≤Week2: number analyzed (Participants) | 63 | 66
  BCSP 4.3-<4.7mEq/L: >Week1 and ≤Week2 | 57 | 57
  BCSP 4.3-<4.7mEq/L: >Week 2 and ≤Week 3: number analyzed (Participants) | 63 | 65
  BCSP 4.3-<4.7mEq/L: >Week 2 and ≤Week 3 | 59 | 63
  BCSP 4.3-<4.7mEq/L: >Week 3 and ≤Week 4: number analyzed (Participants) | 63 | 66
  BCSP 4.3-<4.7mEq/L: >Week 3 and ≤Week 4 | 61 | 60
  BCSP 4.3-<4.7mEq/L: >Week 4 and ≤Week 6: number analyzed (Participants) | 62 | 66
  BCSP 4.3-<4.7mEq/L: >Week 4 and ≤Week 6 | 61 | 61
  BCSP 4.3-<4.7mEq/L: >Week 6 and ≤Week 8: number analyzed (Participants) | 62 | 65
  BCSP 4.3-<4.7mEq/L: >Week 6 and ≤Week 8 | 61 | 58
  BCSP 4.3-<4.7mEq/L: >Week 8 and ≤Week 10: number analyzed (Participants) | 61 | 63
  BCSP 4.3-<4.7mEq/L: >Week 8 and ≤Week 10 | 58 | 58
  BCSP 4.3-<4.7mEq/L: > Week 10 and ≤ Week 12: number analyzed (Participants) | 62 | 64
  BCSP 4.3-<4.7mEq/L: > Week 10 and ≤ Week 12 | 61 | 61
  BCSP 4.7-<5.1 mEq/L: ≤Week 1: number analyzed (Participants) | 83 | 80
  BCSP 4.7-<5.1 mEq/L: ≤Week 1 | 75 | 66
  BCSP 4.7-<5.1mEq/L: >Week 1 and ≤Week 2: number analyzed (Participants) | 84 | 81
  BCSP 4.7-<5.1mEq/L: >Week 1 and ≤Week 2 | 74 | 65
  BCSP 4.7-<5.1mEq/L: >Week 2 and ≤Week 3: number analyzed (Participants) | 83 | 80
  BCSP 4.7-<5.1mEq/L: >Week 2 and ≤Week 3 | 74 | 65
  BCSP 4.7-<5.1mEq/L: >Week 3 and ≤Week 4: number analyzed (Participants) | 82 | 79
  BCSP 4.7-<5.1mEq/L: >Week 3 and ≤Week 4 | 74 | 61
  BCSP 4.7-<5.1 mEq/L: >Week 4 and ≤Week 6: number analyzed (Participants) | 82 | 79
  BCSP 4.7-<5.1 mEq/L: >Week 4 and ≤Week 6 | 79 | 64
  BCSP 4.7-<5.1mEq/L: >Week 6 and ≤Week 8: number analyzed (Participants) | 82 | 77
  BCSP 4.7-<5.1mEq/L: >Week 6 and ≤Week 8 | 74 | 66
  BCSP 4.7-<5.1mEq/L: >Week 8 and ≤Week 10: number analyzed (Participants) | 81 | 75
  BCSP 4.7-<5.1mEq/L: >Week 8 and ≤Week 10 | 72 | 66
  BCSP 4.7-<5.1mEq/L: >Week 10 and ≤Week 12: number analyzed (Participants) | 82 | 76
  BCSP 4.7-<5.1mEq/L: >Week 10 and ≤Week 12 | 80 | 65
  Overall : ≤Week 1: number analyzed (Participants) | 146 | 146
  Overall : ≤Week 1 | 135 | 128
  Overall : > Week 1 and ≤Week 2: number analyzed (Participants) | 147 | 147
  Overall : > Week 1 and ≤Week 2 | 131 | 122
  Overall : >Week 2 and ≤Week 3: number analyzed (Participants) | 146 | 145
  Overall : >Week 2 and ≤Week 3 | 133 | 128
  Overall : >Week 3 and ≤Week 4: number analyzed (Participants) | 145 | 145
  Overall : >Week 3 and ≤Week 4 | 135 | 121
  Overall : >Week 4 and ≤Week 6: number analyzed (Participants) | 144 | 145
  Overall : >Week 4 and ≤Week 6 | 140 | 125
  Overall : >Week 6 and ≤Week 8: number analyzed (Participants) | 144 | 142
  Overall : >Week 6 and ≤Week 8 | 135 | 124
  Overall : >Week 8 and ≤Week 10: number analyzed (Participants) | 142 | 138
  Overall : >Week 8 and ≤Week 10 | 130 | 124
  Overall : >Week 10 and ≤Week 12: number analyzed (Participants) | 144 | 140
  Overall : >Week 10 and ≤Week 12 | 141 | 126

6. Other Pre Specified Outcome: Participants Having Spironolactone Titrations Over Time
Description: The titration was performed according to the following criteria: Spironolactone was increased in cases of hypertension, decreased or stopped in cases of hypotension and maintained if the blood pressure results were adequate
  The symbols > and ≤ included in the row titles are used to indicate the time interval [">Week1 and ≤Week2" meaning from day 8 until day 14 (included)].
Time Frame: From baseline to Week 12
Population: Intent-to-Treat population (ITT): The ITT population included all participants who were randomized and who took at least 1 dose of spironolactone and at least 1 dose of patiromer/placebo.
  Reported results only include the number of participants having spironolactone titrations over time according to the classification defined below.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 147 | 148
Participants
  Up : ≤Week 1 | 0 | 0
  Up : >Week 1 and ≤Week 2: number analyzed (Participants) | 144 | 144
  Up : >Week 1 and ≤Week 2 | 0 | 0
  Up : >Week 2 and ≤Week 3: number analyzed (Participants) | 138 | 136
  Up : >Week 2 and ≤Week 3 | 88 | 77
  Up : >Week 3 and ≤Week 4: number analyzed (Participants) | 136 | 131
  Up : >Week 3 and ≤Week 4 | 27 | 21
  Up : >Week 4 and ≤Week 6: number analyzed (Participants) | 134 | 127
  Up : >Week 4 and ≤Week 6 | 10 | 11
  Up : >Week 6 and ≤Week 8: number analyzed (Participants) | 133 | 117
  Up : >Week 6 and ≤Week 8 | 6 | 6
  Up : >Week 8 and ≤Week 10: number analyzed (Participants) | 128 | 105
  Up : >Week 8 and ≤Week 10 | 6 | 7
  Up : >Week 10 and ≤Week 12: number analyzed (Participants) | 21 | 23
  Up : >Week 10 and ≤Week 12 | 1 | 0
  Down : ≤Week 1 | 1 | 2
  Down : >Week 1 and ≤Week 2: number analyzed (Participants) | 144 | 144
  Down : >Week 1 and ≤Week 2 | 2 | 0
  Down : >Week 2 and ≤Week 3: number analyzed (Participants) | 138 | 136
  Down : >Week 2 and ≤Week 3 | 2 | 2
  Down : >Week 3 and ≤Week 4: number analyzed (Participants) | 136 | 131
  Down : >Week 3 and ≤Week 4 | 6 | 5
  Down : >Week 4 and ≤Week 6: number analyzed (Participants) | 134 | 127
  Down : >Week 4 and ≤Week 6 | 8 | 7
  Down : >Week 6 and ≤Week 8: number analyzed (Participants) | 133 | 117
  Down : >Week 6 and ≤Week 8 | 5 | 8
  Down : >Week 8 and ≤Week 10: number analyzed (Participants) | 128 | 105
  Down : >Week 8 and ≤Week 10 | 4 | 7
  Down : >Week 10 and ≤Week 12: number analyzed (Participants) | 21 | 23
  Down : >Week 10 and ≤Week 12 | 3 | 1

7. Other Pre Specified Outcome: Number of Participants by Spironolactone Dose Prescribed at Each Visit
Description: QD: Once daily
  QOD: Once every other day
Time Frame: From baseline to Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 147 | 148
Participants
  50 mg QD : Baseline | 0 | 0
  50 mg QD : Week 1 | 0 | 0
  50 mg QD : Week 2 | 0 | 0
  50 mg QD : Week 3 | 86 | 76
  50 mg QD : Week 4 | 105 | 94
  50 mg QD : Week 6 | 106 | 96
  50 mg QD : Week 8 | 106 | 85
  50 mg QD : Week 10 | 106 | 80
  25 mg QD : Baseline | 147 | 148
  25 mg QD : Week 1 | 145 | 144
  25 mg QD : Week 2 | 140 | 142
  25 mg QD : Week 3 | 49 | 57
  25 mg QD : Week 4 | 27 | 34
  25 mg QD : Week 6 | 25 | 28
  25 mg QD : Week 8 | 26 | 24
  25 mg QD : Week 10 | 19 | 20
  25 mg QOD : Baseline | 0 | 0
  25 mg QOD : Week 1 | 1 | 2
  25 mg QOD : Week 2 | 3 | 1
  25 mg QOD : Week 3 | 3 | 2
  25 mg QOD : Week 4 | 3 | 3
  25 mg QOD : Week 6 | 2 | 2
  25 mg QOD : Week 8 | 1 | 4
  25 mg QOD : Week 10 | 2 | 4

8. Other Pre Specified Outcome: Shifts in Selected Laboratory Tests From Baseline to End of Treatment
Description: The end of treatment value is defined as the last non-missing value on or prior to the last spironolactone dose date (from End of Treatment - Case report form) + 3 days
  LLN=Lower limit of the normal range. ULN=Upper limit of the normal range. EoT=End of Treatment
Time Frame: From Baseline to End of Treatment, up to 12 weeks.
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 146 | 147
participants
  Magnesium - Baseline Value <LLN : EoT Value<LLN | 9 | 4
  Magnesium - Baseline Value <LLN : EoT Value Normal | 3 | 8
  Magnesium - Baseline Value <LLN : EoT Value >ULN | 0 | 0
  Magnesium - Baseline Value Normal : EoT Value <LLN | 12 | 7
  Magnesium- Baseline Value Normal: EoT Value Normal | 103 | 109
  Magnesium - Baseline Value Normal : EoT Value >ULN | 6 | 10
  Magnesium - Baseline Value >ULN : EoT Value <LLN | 0 | 0
  Magnesium - Baseline Value >ULN : EoT Value Normal | 10 | 6
  Magnesium - Baseline Value >ULN : EoT Value >ULN | 3 | 3
  Phosphate - Baseline Value <LLN : EoT Value <LLN | 0 | 1
  Phosphate - Baseline Value <LLN : EoT Value Normal | 1 | 3
  Phosphate - Baseline Value <LLN : EoT Value >ULN | 0 | 0
  Phosphate - Baseline Value Normal : EoT Value <LLN | 0 | 1
  Phosphate- Baseline Value Normal: EoT Value Normal | 136 | 125
  Phosphate - Baseline Value Normal : EoT Value >ULN | 2 | 8
  Phosphate - Baseline Value >ULN : EoT Value <LLN | 0 | 0
  Phosphate - Baseline Value >ULN : EoT Value Normal | 5 | 4
  Phosphate - Baseline Value >ULN : EoT Value >ULN | 2 | 5
  Calcium - Baseline Value <LLN : EoT Value <LLN | 2 | 4
  Calcium - Baseline Value <LLN : EoT Value Normal | 5 | 1
  Calcium - Baseline Value <LLN : EoT Value >ULN | 0 | 0
  Calcium - Baseline Value Normal : EoT Value <LLN | 4 | 6
  Calcium - Baseline Value Normal : EoT Value Normal | 133 | 133
  Calcium - Baseline Value Normal : EoT Value >ULN | 0 | 0
  Calcium - Baseline Value >ULN : EoT Value <LLN | 0 | 0
  Calcium - Baseline Value >ULN : EoT Value Normal | 2 | 1
  Calcium - Baseline Value >ULN : EoT Value >ULN | 0 | 2

9. Other Pre Specified Outcome: Spironolactone Dose Level at End of 12 Weeks of Study Treatment
Description: Row title:
  Participants not completing 12W of study treatment: Participants who had not completed 12 weeks of study treatment.
Time Frame: 12 Weeks of Study Treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 147 | 148
Participants
  50 mg QD | 102 | 76
  25 mg QD | 22 | 19
  25 mg QOD | 2 | 3
  Participants not completing 12W of study treatment | 21 | 50

10. Post Hoc Outcome: Number of Participants Requiring Additional New Antihypertensive Medications or Increases to Baseline Antihypertensive Medications
Description: Row Titles:
  * AM: Antihypertensive Medication(s)
  * New AM: Participants who required additional new antihypertensive medication(s)
  * Increases to baseline AM: Participants who required increases to baseline antihypertensive medication(s)
  * Addition new (or increase) AM: Participants who required addition of new antihypertensive medication(s) and/or increases to baseline antihypertensive medications
  * At any time during the study: During study
  * While on study medication: On medication
Time Frame: From baseline to Week 12/Early Termination visit
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
Number analyzed (Participants) | 147 | 148
participants
  New AM : At any time during the study | 0 | 3
  New AM : On medication | 0 | 1
  Increases to baseline AM: During study | 0 | 2
  Increases to baseline AM: On medication | 0 | 1
  Addition new (or increases) AM: During study | 0 | 4
  Addition new (or increases) AM : On medication | 0 | 2

ADVERSE EVENTS:
Time Frame: During Treatment Period (12 weeks); until Follow-up Visit 2 weeks after the Week 12 Visit (or Early Termination Visit).
Arm/Group | Group 1 - Patiromer | Group 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/147 | 1/148
Serious Adverse Events (participants affected / at risk) | 1/147 | 4/148
Other Adverse Events (participants affected / at risk) | 47/147 | 48/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Patiromer (N=147) | Group 2 - Placebo (N=148)
Renal failure (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Aortic rupture (Vascular disorders) | 0 | 1
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Patiromer (N=147) | Group 2 - Placebo (N=148)
Diarrhoea (Gastrointestinal disorders) | 9 | 8
Renal impairment (Renal and urinary disorders) | 13 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 13
Headache (Nervous system disorders) | 9 | 11
Hypotension (Vascular disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. No Confidential Information will be disclosed, excluding CT results from Institution
2. No publication shall be initiated by PI until:

   * 18 months after the conclusion of the Study, defined as the locking of the clinical database
   * the publication of a Multicenter Publication (publication of results from all participating sites)
   * written notice from Sponsor that no Multicenter Publication shall ensue
3. PI shall provide a draft of proposed publication for review at least 60 days in advance

DOCUMENTS (2):
  • Study Protocol (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT03071263/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT03071263/SAP_001.pdf